CLINICAL TRIAL: NCT00168207
Title: The Relationship of Single Nucleotide Polymorphisms in the Interleukin-7 Receptor-α Gene to CD4+ Immune Recovery in HIV Infected Patients Who Begin Antiretroviral Treatment With HAART
Brief Title: IL-7 Receptor Polymorphisms and Immune Recovery With HAART
Status: Completed | Type: Observational
Sponsor: The Alfred (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Jennifer Hoy, Professor Jennifer Hoy, The Alfred
Other Study IDs: 112/05
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Plasma, PBMC and DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim is to investigate the hypothesis that IL7-receptor polymorphisms contribute to the differential immune recovery of CD4 + T cells following HAART

DETAILED DESCRIPTION:
AIM: To examine the association between the four haplotypes of IL-7Rα gene and a cohort of HIV infected patients who have commenced HAART with varying CD4+ T lymphocyte responses.

METHODS: IL-7Rα gene SNPs and haplotypes will be measured by constructing DNA pools, and PCR amplification and DNA sequencing. IL-7Rα expression will be examined using constitutive expression of IL-7Rα, IL-7Rα gene expression, and inducible expression of IL7Rα.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years of age
* First antiretroviral regimen composed of HAART as defined by at least three antiretrovirals
* Controlled viremia for a period of at least 12 months following commencement of HAART. Controlled viremia is defined as HIV viral load of ≤ 500 copies/mL on bDNA testing (versions 2 and 3) and <400 copies/ml measured by RT-PCR assay by 6 months treatment.
* CD4 cell count <500 at commencement of HAART
* Measurement of CD4+ cell count on at least 3 time points, in the 12 months post commencement of HAART.

Exclusion Criteria:

* Exclude patients treated for HIV seroconversion illness
* Exclude patients on immunomodulatory therapy such as IL-2, hydroxyurea or prednisolone or who have received an HIV therapeutic vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients on HAART
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2005-05; Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hoy, A/Prof, Study Director — The Alfred; Sharon Lewin, Professor, Principal Investigator — Alfred Hospital, Melbourne, Vic 3004
Locations (1):
- The Alfred Hospital, Commercial Road, Melbourne, Victoria, Australia